CLINICAL TRIAL: NCT02172339
Title: The Pharmacokinetic, Safety and Tolerability of Tiotropium (4.8 mcg, Single i.v. Dose) in Outpatients With Renal Impairment in Comparison to Healthy Subjects (Open Label, Group Comparison, Two-center Study)
Brief Title: The Pharmacokinetic, Safety and Tolerability of Tiotropium in Outpatients With Renal Impairment in Comparison to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205.134
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Tiotropium Bromide

ARMS (1):
- Tiotropium (Experimental): group comparison (healthy, renal impairment)
  Interventions: Drug: Tiotropium, solution ampoules

INTERVENTIONS:
Drug: Tiotropium, solution ampoules

SUMMARY:
Study to investigate pharmacokinetics of a single i.v. dose of tiotropium (4.8 mcg) in patients with renal impairment in comparison to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects:

   1. Subject with normal renal function ( creatinine clearance of 80% of predicted creatinine clearance in healthy volunteers), as confirmed by normal physical examination including vital signs, ECG and laboratory values

      Calculated creatinine clearance (male);

      = ((140 - age(yr)) x (Wt (kg))) / (72 x predicted serum creatinine (mg/dL))

      Calculated creatinine clearance (female);

      = ((140 - age(yr)) x (Wt(kg))) / (85 x predicted serum creatinine (mg/dL))
   2. Subject with impaired renal function must be of age related good health and without clinically significant abnormalities as assessed during the physical examination. Mildly impaired renal patients were defined as those with creatinine clearance of 40 - 80% of predicted creatinine clearance; moderately impaired renal patients were defined as those with creatinine clearance of 10 - 40% of predicted creatinine clearance. Laboratory values of subjects with renal impairment could have been outside the normal range if the deviations were due to the underlying renal disease.
2. Male or female, age between 40 and 70 years with normal body - weight index (+/- 25%, Broca-index)
3. Subjects with normal 12 - lead ECG recording
4. Subjects with normal physical examination
5. Subjects with normal clinical and laboratory tests (except for indicators of renal impairment)
6. Female of child bearing potential must have a negative pregnancy test
7. All subjects must have a negative HIV-Ab test and negative Hepatitis B test
8. All subjects must have a negative drug screening
9. All subjects must sign a written informed consent prior to enrollment

Exclusion Criteria:

1. Subjects with a history of more then moderate alcohol consumption (more than 1 litre of beer per day or the equivalent amount of alcohol in any other alcoholic beverage, approximately 50 g of alcohol per day). 24 hours before dosing and 24 hours post dosing, alcohol was not permitted
2. Present or past participation in a drug detoxification program
3. Smokers
4. Subjects requiring any concomitant medication not compatible with this study
5. Subjects with hypotension (systolic blood pressure less than 100 mmHg, diastolic less than 60 mmHg) or hypertension (systolic blood pressure more than 165 mmHg or diastolic more than 100 mmHg) under adequate medication
6. Subjects who participated in a clinical trial of any other investigational drug within two months prior to the start of this study
7. Pregnant or lactating women or women of child bearing potential not using a medically approved means contraception. (i.e., oral contraceptives, intrauterine devices, diaphragm)
8. Subjects who donated blood within three months prior to the start of the study
9. Subjects with a history of chronic or recurrent convulsive disorders or ongoing hepatic dysfunction
10. Subjects with ongoing acute systemic illness or recovery from acute systemic illness
11. Subjects with a history of cancer within the last five years
12. Subjects with known hypersensitivity to anticholinergic drugs
13. Subjects with known symptomatic prostatic hypertrophy or bladder neck obstruction
14. Subjects with known narrow-angle glaucoma

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1998-04; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC (0-4h) of plasma levels of tiotropium after dosing) | pre-dose, 7, 15 , 20, 25, 35, 45 minutes and 1, 2, 4 and 8 hours after drug administration
Renal clearance of tiotropium (CLren ) | Day 1, 2, 3, 7, 11, 15, 18, 22 and 25 (0-4h, 4-8h), additionally -4 -0 h on day 1
Terminal half-life of tiotropium | pre-dose, 7, 15 , 20, 25, 35, 45 minutes and 1, 2, 4 and 8 hours after drug administration
Urinary excretion (0-4h) of tiotropium, Ae 0-4h | Day 1, 2, 3, 7, 11, 15, 18, 22 and 25 (0-4h, 4-8h), additionally -4 -0 h on day 1

SECONDARY OUTCOMES:
Change from baseline in Pulse Rate (PR) | baseline, day 1, 2, 3, 7,11, 15,18, 22 and 25
Change from baseline in Blood pressure (BP) | baseline, day 1, 2, 3, 7,11, 15,18, 22 and 25
Number of Participants with Serious and Non-Serious Adverse Events | up to day 25
Change from baseline in electrocardiogram (ECG) | baseline, day 1, 2, 7, 15 and 25
Maximum measured concentration of the analyte in plasma (Cmax ) | pre-dose, 7, 15 , 20, 25, 35, 45 minutes and 1, 2, 4 and 8 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | pre-dose, 7, 15 , 20, 25, 35, 45 minutes and 1, 2, 4 and 8 hours after drug administration
Change in FEV1 (Forced expiratory volume in one second) | baseline, day 1, 2, 3, 7,11, 15,18, 22 and 25
Change in FVC (Forced vital capacity) | baseline, day 1, 2, 3, 7,11, 15,18, 22 and 25